CLINICAL TRIAL: NCT01997983
Title: Pilot Study Evaluating Efficacy and Safety of Intravesical Instillations of Botulinum Toxin in TC-3 Gel in Interstitial Cystitis Patients
Brief Title: Efficacy and Safety of Intravesical Instillations of Botulinum Toxin in TC-3 Gel in IC Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-IC-01
Record Dates: First submitted 2013-11-24; First posted 2013-11-28 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Interstitial Cystitis; IC
Keywords: interstitial cystitis; PBS/IC; IC; Botox; Botulinum toxin; TC-3 Gel; TCGel; TheraCoat
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TC-3 Gel with Botox (Experimental): open label observational study
  Interventions: Device: TC-3 Gel mixed with Botox (BTX)

INTERVENTIONS:
Device: TC-3 Gel mixed with Botox (BTX) — TC-3 gel mixed with Botox (BTX). Single intravesical instillations of 40 ml of TC-3 mixed with 200 units of preconstitued BTX, using catheter
  Other Names: botulinum toxin; BTX; TC-3 Gel

SUMMARY:
The investigators believe that this study is of importance of several aspects:

1. It evaluates a new mode of bladder instillation that may bypass the drawbacks of the current instillation mode.
2. It will demonstrating safety of intravesical instillations of BTX mixed with TC-3 gel in IC patients
3. If proved effective or partially effective, this mode of treatment will serve as a basis for large feasibility study exploring its safety and efficacy aspects.

DETAILED DESCRIPTION:
American Urology Association (AUA) considers intradetrusor injection of BTX as a fifth-line treatment of interstitial cystitis due to the seriousness and of adverse events, including dysuria, large post-void residuals, and the need for intermittent self-catheterization. An appealing alternative for BTX injection is intravesical instillation of BTX since the recent studies suggest that intravesically applied BTX acts through the afferent neuropathway involving sensory mechanism in the urothelium rather than the smooth muscle. TheraCoat core technology is based on a reverse thermal biodegradable gel (TC-3) (low viscosity at 5°C gel appearance at body temperature) for drug retention in the urinary bladder. Intravesical BTX instillation using TheraCoat gel is expected to increase treatment efficiency due to prolongation of treatment duration and consequently improving bladder exposure to BTX.

Prior to instillation, the TC-3 hydrogel, in a liquid state, is mixed with BTX.TC-3 mixed with BTX is instilled to the bladder by a catheter. Following gel insertion to the bladder, the gel solidifies and forms a drug reservoir inside the bladder. Upon contact with urine the gel dissolves and is cleared out from the bladder Post instillation, patients followed at 2, 6, 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with Interstitial Cystitis/PBS.
2. Subject has signed Informed Consent Form and is willing and able to abide by the protocol.
3. Subject has IC Symptom index (of IC Symptom and Problem Questionnaire) score of 12-20 points.
4. Subject has IC Problem index (of IC Symptom and Problem Questionnaire) score of 12-16 points.
5. Subject is willing and able to complete the micturition diary and questionnaire correctly.
6. Subject agrees to be available for the follow-up evaluations as required by the protocol.
7. Subject is mentally competent with the ability to understand and comply with the requirements of the study.
8. No active urinary tract infection as confirmed by urine culture.
9. If the subject is a female of childbearing potential she has a negative pregnancy test at screening.

Exclusion Criteria:

1. Patient who is pregnant, lactating, or planning to become pregnant within the study period.
2. Patient used Clean Intermittent Catheterization (CIC).
3. Patient has a known neurological cause for IC/PBS symptoms.
4. Patient has Patient with implanted permanent neuro-stimulation device
5. Patient with pelvic organ prolapse stage III or IV, (i.e. the most distal part of the prolapse protruding more than 1 cm beyond the hymen at straining)
6. Patient with lower tract genitourinary malignancies
7. Patient with prior anti-incontinence surgery and interventions including mid-urethral slings, burch bladder suspension, sacral neuromodulation, or tibial nerve stimulation.
8. Patient received intradetrusor Botox (Botolinum Toxin A) injection within 12 months prior to the study initiation.
9. Patient with previous pelvic radiation therapy
10. Patient who is morbidly obese (BMI > 40 Kg/m2).
11. Patient with current culture-proven urinary tract infection, including cystitis or urethritis.
12. Patient had been treated for 2 or more UTIs within last 6 months.
13. Patient with a life expectancy of less than 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
VAS score | week 12
  Change from baseline in Visual Analog Scale (VAS) score for bladder pain measured at week 12 post BTX+TC-3 instillation.

SECONDARY OUTCOMES:
Number of voids in 24hour period | 12 weeks post instillation
  Change from baseline in number of voids in 24-hour period per 3-day voiding diary measured at week 12 post BTX+TC-3 instillation.
NUmber of urge episodes in 24-hour period | 12 weeks post instillation
  Change from baseline in number of urge episodes in 24-hour period per 3-day voiding diary measured at week 12 post BTX+TC-3 instillation.
number of nocturnal voids in one night | 12 weeks post instillation
  Change from baseline in number of nocturnal voids in one night per 3-day voiding diary measured at week 12 post BTX+TC-3 instillation.
O'Leary-Sant Interstitial Cystitis Symptom index | 12 weeks post instillation
  Change from baseline in O'Leary-Sant Interstitial Cystitis Symptom index per O'Leary-Sant Interstitial Cystitis Symptom and Problem questionnaire measured at week 12 post BTX+TC-3 instillation.

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Zisman, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel